CLINICAL TRIAL: NCT00795405
Title: Cardiovascular Effects of Major Sporting Events in Subjects With Coronary Heart Disease
Brief Title: Cardiovascular Effects of Sporting Events
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Shengshou Hu / President, Cardiovascular Institute & Fuwai Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: sporting events
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Coronary Heart Disease
Keywords: sporting events; stress; myocardial ischemia; ST-segment depression; blood pressure
MeSH Terms: conditions — Coronary Disease; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Sham Comparator): No exposure to sporting events
  Interventions: Behavioral: No exposure to sporting events
- 2 (Experimental): Exposure to sporting events
  Interventions: Behavioral: Exposure to sporting events

INTERVENTIONS:
Behavioral: Exposure to sporting events — Exposure to sporting events
  Arms: 2
Behavioral: No exposure to sporting events — No exposure to sporting events
  Arms: 1

SUMMARY:
Major sporting events may have adverse cardiovascular effects in subjects with coronary heart disease. We also hypothesized that the adverse cardiovascular effects of sporting events are a result of psychobiological processes including stress-induced hemodynamic changes, autonomic dysfunction and parasympathetic withdrawal, and inflammatory and prothrombotic responses, all of which may in turn promote myocardial ischemia.

DETAILED DESCRIPTION:
Observational studies suggest that exposure to sporting events may worsen symptoms of angina and trigger acute myocardial infarction. The mechanisms for this association are unknown. To date, there have been no controlled exposures in patients with coronary heart disease: an important population who may be particularly susceptible to the adverse cardiovascular effects of sporting events.

In a randomized crossover controlled study, 38 patients with prior myocardial infarction will be exposed to sporting events or not. Myocardial ischemia will be quantified by ST-segment analysis using continuous 12-lead electrocardiography, and blood pressure change will be analyzed using ambulatory blood pressure monitoring. Autonomic function will be assessed by heart rate variability. Ischemic, inflammatory and prothrombotic markers will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Previous myocardial infarction (>6 months previously)treated by coronary revascularization
* On standard secondary preventative therapy

Exclusion Criteria:

* Angina pectoris (Canadian Cardiovascular Society grade ≥2)
* History of arrhythmia
* Uncontrolled hypertension
* Unstable coronary disease (acute coronary syndrome or unstable symptoms within 3 months)
* Occupational exposure to sporting events
* Diabetes
* Hepatic or renal failure

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Evidence of definite myocardial ischemia confirmed by Holter monitoring | 2 months
Blood pressure measured by ambulatory blood pressure monitoring | 2 months
Heart rate variability | 2 months

SECONDARY OUTCOMES:
Episode of angina | 3 months
Episode of neurological events | 3 months
Episode of arrhythmia | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Shengshou Hu, MD, Principal Investigator — Cardiovascular Institue and Fuwai Hospital